CLINICAL TRIAL: NCT05070819
Title: Role of Atrial Natriuretic Peptide in Assessing of Fluid Status in Cardiac Surgery Patients
Brief Title: Atrial Natriuretic Peptide in Assessing Fluid Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Petrovsky National Research Centre of Surgery (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0394227092021
Record Dates: First submitted 2021-09-27; First posted 2021-10-07 (Actual); Results first posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Fluid Overload; Fluid Loss; Volume Overload; Cardiac Disease; Cardiac Output, Low; Cardiac Output, High
Keywords: fluid responsiveness; fluid status; cardiac surgery; volemic status; pro-ANP; hemodynamic monitoring; functional test; teboul test; stroke volume variation; cardiac output
MeSH Terms: conditions — Edema; Heart Diseases; Cardiac Output, Low; Cardiac Output, High

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardiac surgery patients (Experimental): 1. After admission to OR and arterial catheter is placed the pro-ANP probe is obtained.
  2. After anesthesia induction, trachea intubation before Teboul' test pro-ANP is obtained
  3. At the end of Teboul' test when lower limbs are lifted
  4. 30 minutes of CPB
  5. End of CPB
  6. End of volume transition from CPB circuit to patient
  7. Before Teboul' test at the end of surgery
  8. End of Teboul' test when lower limbs are lifted
  Interventions: Diagnostic Test: pro-ANP

INTERVENTIONS:
Diagnostic Test: pro-ANP — pro-ANP samples and fluid status assessment with functional tests (Teboul test) will be used 8 times intraoperatively.

SUMMARY:
Biomarkers can play a significant role in fluid status assessment intraoperatively.

DETAILED DESCRIPTION:
Routinely intraoperatively the fluid status assessment is based on central venous pressure and other parameters. Nevertheless, the minority of anesthesiologists use continous dynamic parameters like pulse pressure variation, stroke volume variation and other to manage fluid status. There's a fast acting biomarker that can help anesthesiologist to diagnose and manage the volemic status and possibly guide the infusion therapy better.

Pro-ANP is a biomarker that reacts on atria strain and can be used in volemic status assessment in cardiac surgery patients.

ELIGIBILITY:
Inclusion Criteria:

CABG, one-, two valve repair/replacement, ascending aorta, aortic arch replacement, ASD/AVD closure, septal myectomy

Exclusion Criteria:

1. Atrial fibrillation, atrial flutter, frequent ventricular and supraventricular arrythmias
2. EFLV < 50%
3. Pulmonary hypertension > 2 st
4. CKD > C3 (GFR < 30)
5. Redo surgery
6. Left atrium volume > 150 ml
7. LV EDV > 250 ml

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boris Akselrod, Ph.D, Principal Investigator — Petrovsky NRCS
Locations (1):
- Petrovsky Research National Centre of Surgery (Petrovsky NRCS), Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Influence of volemic status on serum atrial natriuretic peptide in cardiac surgical patients — https://doi.org/10.17116/kardio20231601132

RESULTS

PARTICIPANT FLOW:
Groups:
- Cardiac Surgery Patients: 1. After admission to OR and arterial catheter is placed the pro-ANP probe is obtained.
  2. After anesthesia induction, trachea intubation before Teboul' test pro-ANP is obtained
  3. At the end of Teboul' test when lower limbs are lifted
  4. 30 minutes of CPB
  5. End of CPB
  6. End of volume transition from CPB circuit to patient
  7. Before Teboul' test at the end of surgery
  8. End of Teboul' test when lower limbs are lifted
  pro-ANP: pro-ANP samples and fluid status assessment with functional tests (Teboul test) will be used 8 times intraoperatively.
Period: Overall Study
Arm/Group | Cardiac Surgery Patients
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Cardiac Surgery Patients: 30 patients enrolled in a study
Arm/Group | Cardiac Surgery Patients
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Russia | 30
Body surface area, м² [Mean (Standard Deviation); unit: square meters] | 2 (0.23)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Pro-ANP Twofold Raise by the End of Surgery
Description: To assess the atria strain and consequent rise of pro-ANP by the end of surgery
Time Frame: intraoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Cardiac Surgery Patients
Number analyzed (Participants) | 30
Participants | 17

2. Primary Outcome: Number of Patients With Pro-ANP Increase > 10% by the PLR Maneuver
Description: According to positive PLR the assessment of pro-ANP consequent raise
Time Frame: intraoperative
Measure: Count of Participants; unit: Participants
Groups:
- Cardiac Surgery Patients: At the end of Teboul' test when lower limbs are lifted
Arm/Group | Cardiac Surgery Patients
Number analyzed (Participants) | 30
Participants | 5

3. Primary Outcome: Number of Patients With Cardiac Index Rise > 10% After Passive Leg Raising Maneuver
Description: Using Massimo vigileo hard- and software the first assessment of cardiac index was made before Teboul test after the trachea intubation. After 10 minutes of passive leg raising maneuver second assessment. If raise in cardiac index above 10 percent was detected the patient was considered a responder. If not - non-responder.
Time Frame: 10 minutes of PLR test
Measure: Number; unit: Responders
Groups:
- Cardiac Surgery Patients: Cardiac index assessment at the end of PLR test
Arm/Group | Cardiac Surgery Patients
Number analyzed (Participants) | 30
Responders | 5

4. Primary Outcome: Number of Patients With Pro-ANP Increase > 10% by the PLR Maneuver at the End of Surgery
Description: Using Massimo vigileo hard- and software the assessment of cardiac index was made before Teboul test at the end of surgery before leaving the operating room. After 10 minutes of passive leg raising maneuver second assessment. If raise in cardiac index above 10 percent was detected the patient was considered a responder. If not - non-responder.
Time Frame: 10 minutes of PLR test
Measure: Number; unit: Responders
Groups:
- Cardiac Surgery Patients: End of Teboul' test when lower limbs are lifted
Arm/Group | Cardiac Surgery Patients
Number analyzed (Participants) | 30
Responders | 8

5. Secondary Outcome: Postoperative Complications
Description: Total amount of various postoperative complications
Time Frame: up to 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cardiac Surgery Patients
Number analyzed (Participants) | 30
Participants | 8

6. Secondary Outcome: Mortality
Description: Mortality rate
Time Frame: up to 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cardiac Surgery Patients
Number analyzed (Participants) | 30
Participants | 0

7. Secondary Outcome: Multiorgan Failure
Description: Number of more than 2 organs failure
Time Frame: up to 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cardiac Surgery Patients
Number analyzed (Participants) | 30
Participants | 0

8. Secondary Outcome: Respiratory Failure
Description: Number of patients who require prolonged and/or repeated artificial lung ventilation
Time Frame: up to 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cardiac Surgery Patients
Number analyzed (Participants) | 30
Participants | 0

9. Secondary Outcome: Renal Failure
Description: Number of patients who require extracorporeal detoxication
Time Frame: up to 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cardiac Surgery Patients
Number analyzed (Participants) | 30
Participants | 0

10. Secondary Outcome: Heart Failure
Description: Need in medicamental cardiotonic support more than 1 day
Time Frame: up to 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cardiac Surgery Patients
Number analyzed (Participants) | 30
Participants | 1

11. Secondary Outcome: Circulatory Insufficiency
Description: Need in medicamental vasopressor support more than 1 day
Time Frame: up to 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cardiac Surgery Patients
Number analyzed (Participants) | 30
Participants | 3

12. Secondary Outcome: Infection Rate
Description: Number of patients who develop systemic infection and/or operation wound infection
Time Frame: up to 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Cardiac Surgery Patients
Number analyzed (Participants) | 30
Participants | 0

13. Secondary Outcome: Length of Intensive Care Stay
Description: Duration of summarized length in ICU, including readmission to ICU
Time Frame: up to 10 days
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Cardiac Surgery Patients
Number analyzed (Participants) | 30
hours | 22 [19 to 23]

ADVERSE EVENTS:
Time Frame: 10 days postoperative
Description: All-cause mortality: 0/30
Arm/Group | Cardiac Surgery Patients
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-15): https://cdn.clinicaltrials.gov/large-docs/19/NCT05070819/Prot_SAP_000.pdf